CLINICAL TRIAL: NCT00560430
Title: Regulation of Inflammatory Parameters by Telmisartan in Hypertensive Patients
Acronym: METATEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Bayer (Industry)
Responsible Party: Klaus Parhofer, Principal investigator, Ludwig-Maximilians - University of Munich, Med. Dept. 2,
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: KPUK0106; EudraCT 2006-003567-31
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2010-07-15 (Estimated); Status verified 2008-05

CONDITIONS: Hypertension; Metabolic Syndrome; Hypertriglyceridemia
MeSH Terms: conditions — Hypertension; Metabolic Syndrome; Hypertriglyceridemia | interventions — Telmisartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- T1 (Active Comparator): Telmisartan 80 mg/d
  Interventions: Drug: telmisartan
- T2 (Active Comparator): Telmisartan 160 mg/d
  Interventions: Drug: telmisartan
- P (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: telmisartan — 80 mg per day, orally, weeks 1-14
  Arms: T1
Drug: telmisartan — 80 mg per day; orally, weeks 1 and 2; 160 mg per day; orally, weeks 3-14
  Arms: T2
Drug: placebo — placebo; orally weeks 1-14
  Arms: P

SUMMARY:
A number of studies have shown that certain blood-pressure medications such as ACE-inhibitors and angiotensin-II-receptor blockers (ARB) can reduce the incidence of diabetes mellitus type 2. This protocol will evaluate whether inflammatory mechanisms mediate this effect. The investigators therefore will investigate the effect of telmisartan, a potent ARB, on lipid metabolism, glucose metabolism and inflammation in patients with the metabolic syndrome. Specific parameters will be tested before treatment and after 3 months of treatment. Placebo will be compared to 2 different doses of telmisartan per day.

ELIGIBILITY:
Inclusion Criteria:

* Abd. obesity (BMI>25kg/m²) and waist circumference ≥95cm (men),≥80cm (women)
* Blood pressure ≥130 mmHg (systolic) and/or ≥85 mmHg (diastolic)
* Triglycerides 150-400 mg/dl
* Normal stress test
* Normal carotid ultrasound
* Normal fundoscopy

Exclusion Criteria:

* Diabetes mellitus
* Secondary cause for insulin resistance
* LDL-cholesterol >190 mg/dl
* Atherosclerotic disease
* Blood pressure >160 mmHg (systolic) and/or >100 mmHg (diastolic)
* Regular alcohol consumption (>30 g/day)
* Contraindication against telmisartan
* Antihypertensive medications
* Lipid lowering therapy
* Malignancy
* Pregnancy or Lactation
* Women without adequate contraception

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
change in IL-6 | 14 weeks

SECONDARY OUTCOMES:
change in fasting lipids; | 14 weeks
change in postprandial lipid metabolism | 14 weeks
change in inflammatory parameters | 14 weeks
change in glucose metabolism | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Klaus G Parhofer, MD, Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (2):
- Germany (2):
  - Center for Cardiovascular Research, University Berlin, Berlin
  - Med. Dept. 2, University Munich, Munich